CLINICAL TRIAL: NCT02511145
Title: Exploratory Study to Compare Mechanical Penetration Enhancers on Metvixia Skin Penetration
Brief Title: Comparison of Mechanical Penetration Enhancers on Metvixia Skin Penetration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: RD.03.SPR.40221E; 2013-003371-35 (EudraCT Number)
Record Dates: First submitted 2015-07-28; First posted 2015-07-29 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: volunteers
MeSH Terms: interventions — Occlusive Dressings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Microneedles pretreatment and Metvixia (Active Comparator): minizone with Microneedles pretreatment and Metvixia cream application
  Interventions: Device: Microneedles pretreatment; Drug: METVIXIA Cream
- Microneedles pretreatment and Metvixia under occlusion (Active Comparator): minizone with Microneedles pretreatment and Metvixia cream application with occlusion
  Interventions: Other: occlusive bandage; Device: Microneedles pretreatment; Drug: METVIXIA Cream
- Laser pretreatment and Metvixia (Active Comparator): minizone with laser pretreatment and Metvixia cream application
  Interventions: Device: ablative fractional CO2 laser pretreatment; Drug: METVIXIA Cream
- Laser pretreatment and Metvixia under occlusion (Active Comparator): minizone with Laser pretreatment and Metvixia cream application with occlusion
  Interventions: Other: occlusive bandage; Device: ablative fractional CO2 laser pretreatment; Drug: METVIXIA Cream
- Metvixia (Active Comparator): minizone with Metvixia cream application, without pretreatment
  Interventions: Drug: METVIXIA Cream
- Metvixia under occlusion (Active Comparator): minizone with Metvixia cream application under occlusion, without pretreatment
  Interventions: Other: occlusive bandage; Drug: METVIXIA Cream
- Microneedles pretreatment only (Experimental): minizone with Microneedles pretreatment only
  Interventions: Device: Microneedles pretreatment
- Laser pretreatment only (Experimental): minizone with Laser pretreatment only
  Interventions: Device: ablative fractional CO2 laser pretreatment
- Normal skin (No Intervention): Normal skin control mini-zone

INTERVENTIONS:
Other: occlusive bandage
  Arms: Laser pretreatment and Metvixia under occlusion; Metvixia under occlusion; Microneedles pretreatment and Metvixia under occlusion
Device: ablative fractional CO2 laser pretreatment
  Arms: Laser pretreatment and Metvixia; Laser pretreatment and Metvixia under occlusion; Laser pretreatment only
Device: Microneedles pretreatment
  Other Names: Dermaroller
  Arms: Microneedles pretreatment and Metvixia; Microneedles pretreatment and Metvixia under occlusion; Microneedles pretreatment only
Drug: METVIXIA Cream
  Other Names: MAL
  Arms: Laser pretreatment and Metvixia; Laser pretreatment and Metvixia under occlusion; Metvixia; Metvixia under occlusion; Microneedles pretreatment and Metvixia; Microneedles pretreatment and Metvixia under occlusion

SUMMARY:
Exploratory, mono-center, randomized, intra-individual, controlled trial involving healthy volunteers to compare the effect on MAL penetration into the skin following various mechanical penetration enhancement techniques.

DETAILED DESCRIPTION:
At baseline, each mini-zone was selected and randomly assigned to a pretreatment: 3 zones with microneedling Dermaroller®, 3 zones with ablative fractional CO2 Laser, and 3 zones with no pretreatment. After performing pretreatment, MAL cream was applied on the 6 assigned mini-zones for 3 hours incubation. Each condition was tested with and without occlusion. The three mini-zones with no product applied were used to perform biophysics measures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non childbearing potential, who is at least 18 years of age or older at screening visit.
* The subject has a skin phototype of I to III on Fitzpatrick's scale (Fitzpatrick et al., 1993) at screening visit.
* Subject should have 9 mini zone areas on the back that will be able to receive pre-treatments according to protocol. (checked at Screening visit, and assigned at Baseline visit)
* Female of non childbearing potential (postmenopausal [absence of menstrual bleeding for 1 year prior to screening visit, without any other medical reason], hysterectomy or bilateral oophorectomy).

Exclusion Criteria:

* Subject with porphyria,
* Subject with past history of skin cancer, or current clinical diagnosis of other skin disease (including non-melanoma skin cancer), or tattoos, or cheloid and hypertrophic scars on the test zones, which, in the opinion of the investigator, might interfere with the interpretation of the clinical results,
* Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with the interpretation of the clinical trial results, and/or put the subject at significant risk (according to Investigator's judgment) if he/she participates in the clinical trial.
* Known or suspected allergies or sensitivities to any components of any of the study drugs (see Product label).
* The subject has received, applied or taken some specific treatments within specified time frame prior to the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
fluorescence of protoporphyrin IX (PpIX) | 3 hours